CLINICAL TRIAL: NCT03498287
Title: Randomized Controlled Clinical Trial of Non-invasive Device to Alleviate Carpal Tunnel Syndrome
Brief Title: Non-invasive CTS Device Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pressure Profile Systems, Inc. (Industry)
Collaborators: The Cleveland Clinic (Other); Mission Pain and Spine (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPS-CTS-SBIR2
Record Dates: First submitted 2018-04-08; First posted 2018-04-13 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; carpal tunnel; CTS; musculoskeletal disorder; peripheral neuropathy; repetitive stress injury; non-invasive device; non-significant risk; medical device; wrist pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy; Musculoskeletal Diseases; Peripheral Nervous System Diseases; Cumulative Trauma Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Study Device (Experimental): Small, non-invasive, stiff patch for the wrist
  Interventions: Device: Study Device
- Sham Device (Sham Comparator): Device that looks like the Study Device but modified to prevent or remove the main mechanism of action.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Study Device — Real study device applied to affected wrist (or higher CTS severity wrist if patient has bilateral CTS) for 8-10 hours daily for 56 days (8 weeks).
  Arms: Study Device
Device: Sham Device — Sham device applied to affected wrist (or higher CTS severity wrist if patient has bilateral CTS) for 8-10 hours daily for 56 days (8 weeks). *Note: participants in the sham group are given the real study device at the end of the Post-Treatment/Follow-up Phase.
  Arms: Sham Device

SUMMARY:
Sham-controlled, multi-center and remote patient-centered randomized controlled clinical trial to investigate the efficacy of a novel non-invasive, unobtrusive study device in reducing symptoms of carpal tunnel syndrome (CTS). Daily wear of the study device is expected to significantly reduce symptom severity (evaluated by the Boston Carpal Tunnel Questionnaire) in mild to severe CTS-diagnosed patients. Subjects are randomized into the active device group or sham group for 8 weeks, then followed for 12 weeks post-treatment.

DETAILED DESCRIPTION:
It is hypothesized that daily wear of the study device will result in significant improvements in patient-reported symptom severity. It is also hypothesized that the effects from active study device treatment will be significantly greater than effects from sham treatment. In both cases, it is hypothesized that improvements will be sustained post-treatment.

This study is designed as a randomized, double-blind, sham-controlled, two-arm trial consisting of an eight-week treatment period (active study device or sham), followed by one required follow-up four weeks later (at week 12).

There are two study groups: the active device group receiving the active study device and the sham group receiving a non-active sham device. Subjects will be informed that they have a 50:50 chance of receiving treatment or a sham. They will also be informed that if they receive sham device, they will be offered the active device 4 weeks into the post-treatment period. However, all subjects will not know what treatment they are on until the conclusion of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed with mild to severe carpal tunnel syndrome (CTS)
2. CTS diagnosis confirmed by a nerve conduction study (NCS) performed within the past 24 months OR at enrollment/baseline visit

   1. CTS severity determined via AANEM criteria 13
   2. Bilateral CTS accepted (worse wrist via NCS and/or BCTQ is designated as the study wrist)
3. BCTQ SSS > 2
4. Reliable access to and ability to use Internet, Wi-Fi, or mobile data through computers, mobile devices, laptops, and/or tablets
5. Willing to abstain from any other treatment or therapies for CTS throughout the study
6. Ability to read and write English, or has a reliable person to assist with reading and writing English

Exclusion Criteria:

1. Other upper extremity neuropathies (e.g., epicondylitis, radial nerve neuropathies, ulnar nerve neuropathies)
2. Double crush syndrome
3. Cervical stenosis
4. Brachial plexopathy
5. Wrist fractures or cysts
6. Prior wrist surgeries, especially carpal tunnel release surgery
7. Injection of corticosteroid/cortisone into the wrist or hand within the past 6 months
8. Thyroid disease
9. Rheumatoid arthritis
10. Diabetes
11. Systemic diseases
12. Connective tissue diseases
13. Fibromyalgia or chronic pain syndrome
14. Diabetic neuropathy
15. BMI > 40
16. Participation in other research studies or clinical trials currently or within the past 2 weeks.

To assess eligibility, visit: carpaltunneltrial.com

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae Son, PhD, Study Director — Pressure Profile Systems
Locations (3):
- United States (3):
  - Mission Pain & Spine, Mission Viejo, California
  - South Bay Medical Center, Torrance, California
  - Cleveland Clinic (Lerner Research Institute), Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leite JC, Jerosch-Herold C, Song F. A systematic review of the psychometric properties of the Boston Carpal Tunnel Questionnaire. BMC Musculoskelet Disord. 2006 Oct 20;7:78. doi: 10.1186/1471-2474-7-78. PMID 17054773
- See also: Practice Parameter for Electrodiagnostic Studies in Carpal Tunnel Syndrome: Summary Statement. — http://www.aanem.org/Practice/Guidelines-and-Performance-Measures

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Device: Small, non-invasive, orthodontic arch with adhesive applied to the wrist
  Study Device: Real study device applied to affected wrist (or higher CTS severity wrist if patient has bilateral CTS) for 8-10 hours daily for 56 days (8 weeks). (1 wrist per participant)
- Sham Device: Device that looks like the Study Device but modified to prevent or remove the main mechanism of action.
  Sham Device: Sham device applied to affected wrist (or higher CTS severity wrist if patient has bilateral CTS) for 8-10 hours daily for 56 days (8 weeks). (1 wrist per participant)
  *Note: participants in the sham group were given the real study device at the end of the Post-Treatment/Follow-up Phase.
Period: Overall Study
Arm/Group | Study Device | Sham Device
Started | 45 | 43
Completed | 42 | 38
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Protocol Violation | 0 | 4
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Device: Small, non-invasive, orthodontic arch with adhesive applied to the wrist
  Study Device: Real study device applied to affected wrist (or higher CTS severity wrist if patient has bilateral CTS) for 8-10 hours daily for 56 days (8 weeks).
- Sham Device: Device that looks like the Study Device but modified to prevent or remove the main mechanism of action.
  Sham Device: Sham device applied to affected wrist (or higher CTS severity wrist if patient has bilateral CTS) for 8-10 hours daily for 56 days (8 weeks). *Note: participants in the sham group were given the real study device at the end of the Post-Treatment/Follow-up Phase.
- Total: Total of all reporting groups
Arm/Group | Study Device | Sham Device | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 37 | 79
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (11.7) | 48.6 (9.9) | 48.6 (10.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 34 | 27 | 61
  Male | 8 | 10 | 18
  Decline to Answer | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 25 | 22 | 47
  Unknown or Not Reported | 10 | 13 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 32 | 30 | 62
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 3 | 3 | 6
Boston Carpal Tunnel Questionnaire (BCTQ) Symptom Severity Score (SSS) [Mean (Standard Deviation); unit: units on a 1-5 Likert scale] — enrollment/baseline symptom severity score on the 1-5 Likert scale with 1 being no symptoms and 5 being worst symptoms Population: 80 per-protocol patients analyzed vs total number enrolled
  units on a 1-5 Likert scale | 2.78 (.58) | 2.96 (.42) | 2.87 (.52)
BCTQ Functional Severity Score (FSS) [Mean (Standard Deviation); unit: units on a 1-5 Likert scale] — enrollment/baseline functional severity score on the 1-5 Likert scale with 1 being no symptoms and 5 being worst symptoms Population: 80 per-protocol patients analyzed vs total number enrolled
  units on a 1-5 Likert scale | 2.21 (.72) | 2.39 (.70) | 2.30 (.71)

OUTCOME MEASURES:

1. Primary Outcome: BCTQ SSS at 8 Weeks vs Baseline
Description: The Symptom Severity Scale (SSS) of the Boston Carpal Tunnel Questionnaire (BCTQ) is an 11-question patient-administered survey that rates the severity of the patient's carpal tunnel syndrome-specific symptoms on a scale of 1 (no symptoms) to 5 (worst symptoms).
Time Frame: baseline and 8 weeks post-Baseline
Population: Per-protocol population (patients that completed at least up to the first post-treatment follow-up (Week 12))
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Device | Sham Device
Number analyzed (Participants) | 42 | 38
score on a scale
  Average SSS | 2.16 (.65) | 2.32 (.70)
  Average Change in SSS | -0.62 (0.69) | -0.64 (0.62)

2. Secondary Outcome: BCTQ SSS
Description: as for outcome 1
Time Frame: 8-weeks post-Baseline and 12 weeks post-Baseline
Population: Per-protocol population (patients that completed at least up to the first post-treatment follow-up (Week 12))
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Device | Sham Device
Number analyzed (Participants) | 42 | 38
score on a scale
  Average SSS @12 weeks | 2.24 (.70) | 2.44 (.68)
  Average Change in SSS between 12 and 8 weeks | 0.08 (0.48) | 0.12 (0.40)

ADVERSE EVENTS:
Time Frame: Patient participation duration: 5-6 months
Description: Device is a non-invasive externally-worn orthotic made of hypoallergenic materials and does not introduce any medications, chemicals, biologics, or electromagnetic energy into the body. Only expected adverse events are related to skin reaction, rash, allergy, discomfort from device wear, and progression of carpal tunnel syndrome.
Arm/Group | Study Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/38
Other Adverse Events (participants affected / at risk) | 2/42 | 2/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study Device (N=42) | Sham Device (N=38)
Rash, redness, or sore under study device (Injury, poisoning and procedural complications) | 2 | 2

LIMITATIONS AND CAVEATS:
Sham device was not thoroughly tested before the trial. Post-trial testing suggest some mechanical effect that could have influenced the sham group response. Early termination of enrollment reduced the power of the statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship will reflect joint cooperation between PPS and participating PI(s). Authorship responsibilities should be established prior to the writing of any manuscript.

No individual publications are allowed unless agreed upon, reviewed, and approved by the Sponsor before submission and/or publication. No individual publications are allowed prior to the completion of a final report for the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03498287/Prot_SAP_001.pdf